CLINICAL TRIAL: NCT00635531
Title: A Randomized, Double-blind, Placebo-controlled Study of Xanax XR in the Treatment of Adolescents With a Primary Diagnosis of Panic Disorder
Brief Title: A Study to Evaluate the Use of Extended Release Alprazolam in the Treatment of Adolescents With Panic Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6131002
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Other: placebo
- Alprazolam XR group (Active Comparator)
  Interventions: Drug: alprazolam XR

INTERVENTIONS:
Other: placebo — Placebo dosing same as alprazolam, except a placebo equivalent was substituted for alprazolam
  Arms: Placebo group
Drug: alprazolam XR — Oral treatment started at a daily dose of 1 mg tablets for the first 7 days; thereafter the daily dosage was titrated at a maximum rate of 1 mg every 7 days up to a maximum dosage of 6 mg for lack of response, and in the absence of dose-limiting adverse events; no further increases in daily dose were permitted after Day 36; dosage reductions were permitted if required for tolerability; subjects who were not eligible for entry into the 18-week continuation study, or who were eligible but elected not to participate, were tapered off study drug at a rate of 1 mg every 7 days for up to a 6-week taper period.
  Other Names: Xanax XR
  Arms: Alprazolam XR group

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, and pharmacokinetics of alprazolam extended release (XR) for the treatment of adolescents with panic disorder

DETAILED DESCRIPTION:
Due to recruitment difficulties in this adolescent population, the clinical program for alprazolam XR was cancelled and this study was terminated on 1 September 2004. There were no safety concerns that led to this decision.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-IV-TR diagnosis of panic disorder with or without agoraphobia based on the Mini International Neuropsychiatric Interview for Children and Adolescents
* At least an average of one 4-symptom panic attack per week over the last 4 weeks prior to screening
* At least an average of one 4-symptom panic attack per week over the last 4 weeks prior to baseline
* At least one 4-symptom panic attack in the 7 days prior to baseline

Exclusion Criteria:

* Current (in the past 6 months) DSM-IV-TR diagnosis of obsessive compulsive disorder, major depressive disorder, dysthymic disorder, or alcohol and/or substance dependence
* Primary DSM-IV-TR diagnosis of social anxiety disorder, post-traumatic stress disorder, simple phobia, separation anxiety disorder, generalized anxiety disorder, conduct disorder, oppositional defiant disorder, or attention deficit hyperactivity disorder
* Any current or past history of schizophrenia or psychosis; bipolar disorder or cyclothymia; dementia, delirium or other organic brain disease; an Axis I eating disorder; mental retardation, Asperger's disorder, or any other serious developmental disorder
* A CDRS-R score >35

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2004-04; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Endpoint change from baseline in the Panic Disorder Severity Scale for Adolescents (PDSS-A) total score | Week 6
Endpoint change from baseline in the weekly frequency of 4-symptom panic attacks | Week 6

SECONDARY OUTCOMES:
Weekly change in the PDSS-A total score | Weeks 1, 2, 3, 4, 5, and 6
Weekly change and endpoint change from baseline in Clinical Global Impression (CGI)-Severity scale | Weeks 1, 2, 3, 4, 5, and 6
Weekly change and endpoint change from baseline in CGI-lmprovement scale | Weeks 1, 2, 3, 4, 5, and 6
Weekly change and and endpoint change from baseline in PDSS-A item scores | Weeks 1, 2, 3, 4, 5, and 6
Endpoint change from baseline in the Hamilton anxiety rating scale total score | Week 6
Endpoint change from baseline in the Children's Depression Rating Scale (CDRS-R) total score | Week 6
Endpoint change from baseline in Pediatric Quality of Life, Enjoyment, Satisfaction Questionnaire | Week 6
Safety assessments will include physical examination, electrocardiogram and laboratory assessments obtained at initial screening, and at the end-of-study visit | Baseline and Week 6
Cognitive and memory effects (free verbal recall test and Digit- Symbol Coding Test) | Baseline and Week 6
Population pharmacokinetic analysis | Weeks 2, 4, and 6
Vital signs | Weeks 1, 2, 3, 4, 5, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Middleton, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131002&StudyName=A%20Study%20to%20Evaluate%20the%20Use%20of%20Extended%20Release%20Alprazolam%20in%20the%20Treatment%20of%20Adolescents%20with%20Panic%20Disorder%20